CLINICAL TRIAL: NCT02248636
Title: Cholinesterase Inhibitor Discontinuation
Acronym: CID
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-014-13F
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Dementia
Keywords: Alzheimer's disease; Cholinesterase inhibitor; Discontinuation
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Cholinesterase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Real discontinuation (Experimental): This group is tapered off their previous cholinesterase inhibitor medication.
  Interventions: Drug: Cholinesterase inhibitor
- Sham discontinuation (Sham Comparator): This group receives their previous cholinesterase inhibitor medication, but in in placebo form.
  Interventions: Drug: Sham discontinuation

INTERVENTIONS:
Drug: Cholinesterase inhibitor — This group receives a half-dose of their previous cholinesterase inhibitor medication (in overencapsulated form) for two weeks, then receives placebo.
  Arms: Real discontinuation
Drug: Sham discontinuation — This group receives their previous dose of cholinesterase inhibitor medication, but in overencapsulated form
  Arms: Sham discontinuation

SUMMARY:
This study tries to determine if stopping certain medications that are used to treat dementia will cause worsening from the patient and family perspective.

All of the participants will take pills that look identical, and that may contain active drug or an inactive pill (a placebo). Half of the group will receive the same treatment they were taking before the study -- this is called the "sham discontinuation" arm. The other half will receive a reduced dose of their medication, and then an inactive pill (placebo) -- this is called the "real discontinuation" arm.

Participants will be able to return to their previous dose of medication at any time during the study. The percentage of people who return will be measured and compared. Other medical events and factors such as behaviors, thinking, and caregiver distress, will be measured and compared between the groups.

DETAILED DESCRIPTION:
There are no reliable findings from controlled trials about discontinuation of cholinesterase inhibitors from a patient and family perspective. It is unknown at what point these medications do not have effects, and how they can safely be discontinued.

The investigators will identify Veterans who have been taking a cholinesterase inhibitor (CI) (donepezil or galantamine) for at least one year. After informed consent, the investigators will randomize them to Real Taper (half-dose of the CI they had taken for 3 weeks, then placebo for 3 weeks), or Sham Taper (continued full dose of the CI they had taken for 6 weeks). The pills will be blinded by over-encapsulating of the drug or placebo.

An intake interview will ascertain history and measure behaviors, cognitive symptoms, and mood, as well as caregiver burden. Phone calls will assess treatment use and adverse events at week 2 and week 4. An exit interview at week 6 will measure the same variables as at baseline. Participants will be unblinded at that point so they will know which treatment had been used. A follow-up call at 12 weeks will ascertain ongoing treatment and any further adverse events.

At any point in the study, participants and caregivers will be able to return to their pre-study dose of medication.

The primary outcome is the percentage of participants who successfully complete a 6-week discontinuation. This will be compared between arms. Other outcomes related to medical events (e.g. hospitalizations, falls), symptoms (e.g. cognition, behaviors), and caregiver distress will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 60 and older.
* Taking stable dose of donepezil 10mg or greater per day, or galantamine 8mg or greater per day, for at least 1 year.
* Presence of a primary caregiver who can assume responsibility for medication compliance, OR residence in a nursing home with a staff member who can provide information.
* Primary care visit within last 12 months.
* Willing to have the CI medication discontinued.

Exclusion Criteria:

* Terminal medical condition for which life expectancy would be less than 6 months.
* Parkinson's Disease
* Presence of any uncontrolled systemic illness that would interfere with participation in the study.
* Unstable medical condition.
* Receiving services from hospice.
* Current prescription with more than one CI
* Receiving medication in an investigational drug study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Thielke, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (4):
- United States (4):
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - Boise VA Medical Center, Boise, ID, Boise, Idaho
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans who have received a prescription for a cholinesterase inhibitor for one year or greater.
Pre-assignment Details: 72 people were enrolled and consented, but only 61 were randomized.
Period: Overall Study
Arm/Group | Real Discontinuation | Sham Discontinuation
Started | 26 | 35
Completed | 20 | 32
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real Discontinuation | Sham Discontinuation | Total
Number analyzed (Participants) | 26 | 35 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 23 | 33 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.34 (10.48) | 77.94 (9.72) | 77.69 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 25 | 35 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 34 | 60
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 25 | 29 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Successful Completion
Description: Participants can return to their pre-study dose of medication at any time. If they complete 6 weeks of either real discontinuation or sham discontinuation, they are considered to have successfully completed treatment.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Real Discontinuation | Sham Discontinuation
Number analyzed (Participants) | 26 | 35
Participants | 20 | 32

2. Secondary Outcome: Caregiver Burden
Description: The Zarit Caregiver Burden Interview contains 22 items, each on a 5-point scale, for a maximum score of 110. The minimum score is 0. A higher score indicates worse subjective burden.
Time Frame: 6 weeks
Population: Not all of the caregivers completed the instrument. Some were unavailable after study enrollment. Some had a change in caregiver. Some refused to respond to all of the questions, since the instrument is rather lengthy.
Measure: Mean (Standard Deviation); unit: Change in Zarit score
Arm/Group | Real Discontinuation | Sham Discontinuation
Number analyzed (Participants) | 12 | 18
Change in Zarit score | 5.58 (11.13) | 1.66 (17.56)

3. Secondary Outcome: Veteran Cognition
Description: Six-Item Screener is a telephone-based assessment of cognitive status. The score ranges from 0 to 6. A higher score indicates better cognition.
Time Frame: 6 weeks
Population: Some of the participants refused to complete the cognitive instrument over the phone.
Measure: Mean (Standard Deviation); unit: Change in Six-Item Screener Score
Arm/Group | Real Discontinuation | Sham Discontinuation
Number analyzed (Participants) | 20 | 30
Change in Six-Item Screener Score | -0.15 (2.13) | 0.13 (0.90)

4. Secondary Outcome: Veteran Functioning
Description: The Alzheimer's Disease Cooperative Study ADL Scale (ADCS-ADL) is a 23-item scale divided into activities of daily living and independent activities of daily living. Scores range from 0-78. A lower score indicates worse functional ability.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real Discontinuation | Sham Discontinuation
Number analyzed (Participants) | 26 | 35
score on a scale | -1.44 (11.87) | -0.59 (6.72)

5. Secondary Outcome: Behavioral Symptoms
Description: The Behavioral Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD) is a 25-item instrument. Scores range from 0-75, with a higher number indicating worse behavioral symptoms.
Time Frame: 6 weeks
Population: Not all caregivers were willing to respond to all the items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real Discontinuation | Sham Discontinuation
Number analyzed (Participants) | 24 | 35
score on a scale | -1.63 (6.26) | -1.23 (3.79)

6. Secondary Outcome: Post-study Treatment Choice
Description: Veteran and caregiver decision to continue, or to have restarted, the pre-study medication at 12 weeks. The participants were unblinded at 6 weeks, and were requested to make their own decision about restarting.
Time Frame: 12 weeks
Population: We were unable to reach some participants at 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Real Discontinuation | Sham Discontinuation
Number analyzed (Participants) | 25 | 32
Participants
  Participants taking pre-study medication | 13 | 25
  Participants not taking pre-study medication | 12 | 7

ADVERSE EVENTS:
Time Frame: Six weeks.
Description: Dementia patients have a variety of behavioral and health events, which may fluctuate over time. We considered adverse events to be novel medical events differing from baseline.
Arm/Group | Real Discontinuation | Sham Discontinuation
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/35
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/35
Other Adverse Events (participants affected / at risk) | 9/26 | 3/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Discontinuation (N=26) | Sham Discontinuation (N=35)
Behavior (Psychiatric disorders) | 9 (9) | 3 (3) — Behavior changed significantly

LIMITATIONS AND CAVEATS:
The study was designed to allow participants to stop the study medication at any time, and for any reason. This is different than administrative withdrawal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT02248636/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT02248636/SAP_001.pdf